CLINICAL TRIAL: NCT00347971
Title: Phase 1, Open-Label, Dose-Escalation Study to Assess the Safety and Pharmacokinetics of Recombinant Interleukin 21 (rIL-21) Administered in Combination With Rituxan (Rituximab) in Subjects With B-Cell Non Hodgkin's Lymphoma
Brief Title: Study of Recombinant Interleukin 21 in Combination With Rituxan for Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ZymoGenetics (Industry)
Responsible Party: Muriel Siadak, ZymoGenetics
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 494E03
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2008-09-05 (Estimated); Status verified 2008-09

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: Lymphoma, Non-Hodgkin; interleukin-21; rituximab; Immunotherapy
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab

INTERVENTIONS:
Drug: recombinant human interleukin 21 and rituximab — rIL-21 (30, 100, 150 ug/kg) IV rituximab (375 mg/m2) IV
  Other Names: rituxan

SUMMARY:
The purpose of the study is to evaluate whether recombinant IL-21 used in combination with rituximab is safe for patients with non-Hodgkin's lymphoma (NHL).

DETAILED DESCRIPTION:
This is a Phase 1 open-label dose-escalation study of rituximab + rIL-21 combination therapy, administered once weekly for 4 weeks following an initial treatment with one dose of rituximab alone to patients with B-cell non-Hodgkin's lymphoma (NHL) who have failed prior therapy(ies). A standard dose of rituximab will be used. Increasing doses of rIL-21 will be studied sequentially in different groups of patients, starting with 30 μg/kg.

Before starting treatment with rituximab + rIL-21, patients will be treated with one dose of rituximab alone to look for rituximab infusion-related symptoms (such as fever, chills, and rigors). Patients who have severe infusion-related side effects after the first dose of rituximab will not go on to receive IL-21. Those who do not have unacceptable rituximab-related side effects will receive intravenous rIL-21 at least 60 minutes after completing the rituximab infusion at the rest of the weekly dosing visits. Patients will be evaluated for safety over the course of the study. Disease evaluation (tumor restaging) will be performed 2 weeks following completion of the first 4-week treatment cycle. Patients with stable disease or better at this evaluation may go on to receive a second 4-week treatment cycle of rituximab + rIL-21. Patients may be in the study for 2 to 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CD20+ B-cell NHL
* Disease measurable by computed tomography (CT) scan
* Has failed at least one prior systemic therapy for NHL
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate hepatic and renal function
* Adequate bone marrow function

Exclusion Criteria:

* Presence of acute infection or other significant systemic illness
* White blood cell (WBC) count > 50,000/mm3 in peripheral blood
* Central nervous system involvement by malignancy
* Previous allogenic transplant or autotransplant within 6 months of enrollment
* Other current malignancy or known history of cancer within 5 years
* Received systemic corticosteroids, chemotherapy, immunotherapy, biologic therapy, antibody therapy (e.g., rituximab), radiation therapy, and/or investigational agent(s) within 1 month of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2006-06; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events through 1 month after completing treatment | During treatment and through 1 month after completing treatment
Incidence and grade of clinical laboratory abnormalities through 1 month after treatment | During treatment and through 1 month after completing treatment

SECONDARY OUTCOMES:
Disease response by the International Workshop to Standardize Response Criteria for Non-Hodgkin's Lymphomas 2 weeks after completion of the first treatment cycle | Two and four weeks after completion of the first and second cycles, respectively
Immunogenicity by incidence of anti-rIL-21 antibodies up to 1 month after treatment | During treatment and up to 1 month after completing treatment

CONTACTS AND LOCATIONS:
Overall Officials: Muriel Siadak, PA-C, Study Director — ZymoGenetics
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States